CLINICAL TRIAL: NCT02856022
Title: A Comparison of the Efficacy of Electrical Ilioinguinal Nerve Stimulation and Intravesical Irrigation in Treating Patients With Bladder Pain Syndrome in Women
Brief Title: A Comparison of Electrical Ilioinguinal Nerve Stimulation With Intravesical Irrigation for Bladder Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Institute of Acupuncture, Moxibustion and Meridian (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZYY201606
Record Dates: First submitted 2016-08-02; First posted 2016-08-04 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2016-06

CONDITIONS: Painful Bladder Syndrome
Keywords: electrical ilioinguinal nerve stimulation; bladder pain syndrome; intravesical irrigation
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electrical ilioinguinal nerve stimulation (Experimental)
  Interventions: Device: Electrical ilioinguinal nerve stimulation
- Intravesical Irrigation (Active Comparator)
  Interventions: Procedure: Intravesical Irrigation

INTERVENTIONS:
Device: Electrical ilioinguinal nerve stimulation — Four abdominal points are selected. The upper two points are located 2.5 cun bilateral to Guanyuan (Ren 4). The lower two points are located 1.5 cun bilateral to Zhongji (Ren 3). Four long needles are punctured obliquely 1~2 cun in depth (depending on the fat layer thickness of the patient) to the four points to make the needling sensation reaching the urethra or vulva.
  After the needling sensation reach the above regions, each of two pairs of electrodes from a device are connected with the two ipsilaterally inserted needles. The parameters are continuous waves, a frequency of 2.5 Hz and intensity that the patient feels comfortable for 60 min, three times a week for at least four weeks.
  Arms: Electrical ilioinguinal nerve stimulation
Procedure: Intravesical Irrigation — The patient was asked to lie on a couch in a lithotomy position after urination. A catheter was passed through the urethra into the bladder and any residual urine drained. The Cystistat 50mL 40mg (sodium hyaluronate, Bioniche Teoranta, Ireland) solution is instilled through the catheter into the bladder. The catheter is then withdrawn leaving the Cystistat inside the bladder coating the lining. It was recommended the solution was retained for as long as possible, ideally at least 30 minutes. The instillation is once weekly for at least four weeks.
  Arms: Intravesical Irrigation

SUMMARY:
The purpose of this study is to determine whether electrical ilioinguinal nerve stimulation (EINS) is more effective than intravesical irrigation (II) in treating bladder pain syndrome.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether electrical ilioinguinal nerve stimulation (EINS) is more effective than intravesical irrigation (II) in treating bladder pain syndrome.

ELIGIBILITY:
Diagnostic Criteria:

1. Complaint of suprapubic pain related to bladder filling, accompanied by other symptoms such as increased daytime and night-time frequency, in the absence of proven urinary infection or other obvious pathology.
2. Negative in urine routine test or urine cultivation.
3. Urinating at least 7 times per day or having some urgency or pain (measured on linear analog scales)

Inclusion Criteria:

1. Providing informed consent to participate in the study;
2. Willing to undergo a cystoscopy under general or regional anesthesia when indicated during the course of the study;
3. Female patients meeting the diagnostic criteria;
4. Age ≥18 years and ≤80 years.
5. Disease course ≥ 6 months

Exclusion Criteria:

1. Bladder capacity of greater than 350 mL on awake cystometry;
2. Absence of an intense urge to void with the bladder is filled to 150 mL of liquid filling medium;
3. The demonstration of phasic involuntary bladder contractions on cystometry using the fill rate just described;
4. Duration of symptoms less than 9 months;
5. Absence of nocturia;
6. Symptoms relieved by antimicrobial agents, urinary antiseptic agents, anticholinergic agents, or antispasmodic agents;
7. A frequency of urination while awake of less than 8 times per day;
8. A diagnosis of bacterial cystitis or prostatitis within a 3-month period;
9. Bladder or ureteral calculi;
10. Active genital herpes;
11. Uterine, cervical, vaginal, or urethral cancer;
12. Urethral diverticulum;
13. Cyclophosphamide or any type of chemical cystitis;
14. Tuberculous cystitis;
15. Radiation cystitis;
16. Benign or malignant bladder tumors;
17. Vaginitis;
18. Age younger than 18 years.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Bladder Pain/ Interstitial Cystitis Symptom Score (BPIC-SS) | 4 weeks

SECONDARY OUTCOMES:
SF-36 questionnaire | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Siyou Wang, M.D, Study Director — Shanghai research institute of acupuncture and meridian
Locations (1):
- Shanghai research institute of acupuncture and meridian, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided